CLINICAL TRIAL: NCT03440138
Title: Defining Benchmarks in Bariatric Surgery - A Global Analysis of Laparoscopic Roux-en-Y Gastric Bypass and Sleeve Gastrectomy
Brief Title: Defining Benchmarks in Bariatric Surgery
Acronym: BBenchmarks
Status: Completed | Type: Observational
Sponsor: Marco Bueter (Other)
Collaborators: Dr. med. Daniel Gero (Unknown); Dr. med. Dimitri A. Raptis, PhD (Unknown); Dr. med. Henner Schmidt (Unknown)
Responsible Party: Sponsor-Investigator, Marco Bueter, Prof. Dr. med., PhD, University of Zurich
Organization: University of Zurich (Other)
Other Study IDs: BASECnr_2017-01652
Record Dates: First submitted 2018-02-07; First posted 2018-02-20 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Benchmark; Bariatric Surgery; Roux-en-y Gastric Bypass; Sleeve Gastrectomy; Complications
MeSH Terms: interventions — Bariatric Surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (19):
- University Hospital Zurich
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- St Pierre University Hospital, Brussels, Belgium
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Sana Klinikum, Offenbach, Germany
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Complutense University of Madrid, Spain
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Musgrove Park Hospital, Taunton, UK
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- University of Gothenburg, Sweden
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- AZ Sint-Jan Hospital in Bruges, Belgium
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Bristol
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Cleveland Clinic, Weston, Florida, USA
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Oswaldo Cruz German Hospital, Sao Paolo, Brazil
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Clínica Las Condes, Santiago, Chile
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Brown University, Providence Rhode Island
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Fresno Bariatric, CA, USA
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Rijnstate Hospital, Arnhem, The Netherlands
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- CHU Nice, France
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Claraspital Basel, Switzerland
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Gastro-Obeso-Center Advanced Med Inst, Brazil
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Hospital Dipreca Santiago Región Metropolitana , Chile
  Interventions: Procedure: bariatric surgery (RYGB or SG)
- Medical University Wien, Austria
  Interventions: Procedure: bariatric surgery (RYGB or SG)

INTERVENTIONS:
Procedure: bariatric surgery (RYGB or SG) — laparoscopic Roux-en-Y gastric bypass or sleeve gastrectomy for severe obesity

SUMMARY:
Aim: To define benchmark outcomes in minimally-invasive primary bariatric surgery.

Design: Multicenter retrospective cohort study.

Assessed outcomes: Morbidity as defined by the Clavien-Dindo classification for surgical complications, the Comprehensive Complication Index® (CCI®) at discharge, at 3 months and at latest follow-up. Evolution of body mass index (BMI) will be also analyzed.

Hospital eligibility: High volume centers (> 200 bariatric operations per year) from at least three continents, maintaining a prospective database, as well as having published previously critically on their outcome.

Study population: Adult patients who underwent primary minimally invasive (laparoscopic / robotic) Roux-en-Y gastric bypass or sleeve gastrectomy from 1st of June 2012 to 31st of May 2017.

Patient Exclusion criteria: detailed later.

Data collection Deadline: 1st September 2017 - 30 April 2018

DETAILED DESCRIPTION:
Background With the growing complexity and cost of modern surgical practice, quality assessment becomes mandatory. The notion of quality and quality assessment is widely recognized and used in the world of business and manufacturing. A possible tool of quality assessment is benchmarking. Benchmarking is a process of measuring performance by comparison to the outcomes achieved by the best "service provider" in a specific domain. Usually, a benchmark describes the ''best possible'' outcome of a benchmarking subject to whom comparison can be performed. In the surgical community, however, such benchmarks - best possible outcomes - for specific procedures, not just the pooled overall performance, are lacking.

In 2016, a first landmark study defining benchmark outcomes for liver resection was published in Annals of Surgery by a group of international authors invited and guided by our department. More recently, further surgical outcomes (liver transplantation, minimally invasive esophagectomy) have been benchmarked and have been accepted for publication.

Since laparoscopic bariatric surgery has become a standardized and widely performed procedure worldwide, quality assessment is of major importance. To identify the best possible outcomes (i.e. the benchmarks), data from high-volume centers (based on official IFSO criteria) in low risk patients will be analyzed. These benchmarks will serve as "optimal outcomes" for comparison with single center outcomes, high-risk patients and future developments.

Aim The primary aim is to define benchmark outcomes based on assessment of post procedural complications according to the Clavien-Dindo classification for surgical complications and the comprehensive complication index CCI™ at discharge and at 90-days. The CCI® expresses morbidity on a continuous numeric scale from 0 (no complications) to 100 (death) by weighing all postoperative complications according to the Clavien-Dindo classification for their respective severity. Secondary outcome measure are patient survival and excess BMI loss (EBMIL).

Data Security This multicenter international study is designed to harvest prospectively collected retrospective data via an encrypted (i.e. Secure Sockets Layer (SSL) protocol) online platform (https://bbenchmarks.org/) that meets Food and Drug Administration (FDA) standards and is accessible only by secured login membership.

Confidential center specific data: Centers' outcomes will be individually analyzed in a first step to screen for center-specific differences. Benchmarks will be computed from each center's results in a second step. No center-specific data will be published. Instead, all complications or adverse outcomes will be anonymously reported, as fractions of the total study population. Each center, of course, will be free to publish their own data, as they wish.

Further use of cohort data: Future studies based on the collected data may emerge from this multicenter study, such as comparing outcomes in patients with or without specific comorbidities with benchmark outcomes. For further data usage, additional ethics approval may be required.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of 18-65 years
* Low risk profile (please read "exclusion criteria"),
* Maximum preoperative BMI of 50 kg/m2
* Primary laparoscopic/robotic proximal Roux-en-Y gastric bypass or sleeve gastrectomy
* Documented follow-up of at least 90 days

Exclusion Criteria:

* Open surgery
* Previous intra-abdominal surgery (including previous bariatric surgery)
* Pre-operative BMI over 50 kg/m2
* Age over 65 years
* Cardiovascular disease (e.g. cardiac arrhythmia, stroke, coronary artery disease) (Hypertension is allowed)
* History of thromboembolic events and/or therapeutic anticoagulation
* Diabetes mellitus (Type I and Type II, as defined by the American Diabetes Association)
* Obstructive sleep apnea (recurrent episodes of upper airway collapse during sleep)
* Chronic obstructive pulmonary disease (FEV1/FVC<0.7)
* Chronic kidney disease (eGFR < 30ml/min/1.72 m2)
* Inflammatory bowel disease (ulcerative colitis, Crohn's)
* Immunosuppression therapy (e.g. steroids, calcineurin inhibitors, etc)
* Patients who underwent associated procedures (for example: cholecystectomy, hiatoplasty, liver biopsy)
* ASA score > 2

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with severe obesity with a lower risk profile who undergo bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 5741 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2018-09-10 (Actual); Study Completion 2019-09-17 (Actual)

PRIMARY OUTCOMES:
Benchmark outcomes (best achievable outcomes after bariatric surgery) | 30 days postoperatively
  Comprehensive Complication Index (http://www.assessurgery.com/calculator_single/)
Benchmark outcomes (best achievable outcomes after bariatric surgery) | 90 days postoperatively
  Comprehensive Complication Index (http://www.assessurgery.com/calculator_single/)
Benchmark outcomes (best achievable outcomes after bariatric surgery) | 180 days postoperatively
  Comprehensive Complication Index (http://www.assessurgery.com/calculator_single/)
Major complications after bariatric surgery | 30 days postoperatively
  Clavien-Dindo grade > IIIa
Major complications after bariatric surgery | 90 days postoperatively
  Clavien-Dindo grade > IIIa
Major complications after bariatric surgery | 180 days postoperatively
  Clavien-Dindo grade > IIIa

SECONDARY OUTCOMES:
Case-mix within centers | 5 years
  proportion of benchmark cases
Excess weight loss after bariatric surgery | 1-year postoperatively
  Body-mass index (kg/m2)
Excess weight loss after bariatric surgery | 3-years postoperatively
  Body-mass index (kg/m2)
Excess weight loss after bariatric surgery | 5-years postoperatively
  Body-mass index (kg/m2)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
the study is based on de-anonymised data, so it is impossible to backtrack it to a patient. only overall data will be shared, not individual data

REFERENCES:
- [Background] Rossler F, Sapisochin G, Song G, Lin YH, Simpson MA, Hasegawa K, Laurenzi A, Sanchez Cabus S, Nunez MI, Gatti A, Beltrame MC, Slankamenac K, Greig PD, Lee SG, Chen CL, Grant DR, Pomfret EA, Kokudo N, Cherqui D, Olthoff KM, Shaked A, Garcia-Valdecasas JC, Lerut J, Troisi RI, De Santibanes M, Petrowsky H, Puhan MA, Clavien PA. Defining Benchmarks for Major Liver Surgery: A multicenter Analysis of 5202 Living Liver Donors. Ann Surg. 2016 Sep;264(3):492-500. doi: 10.1097/SLA.0000000000001849. PMID 27433909
- [Background] Muller X, Marcon F, Sapisochin G, Marquez M, Dondero F, Rayar M, Doyle MMB, Callans L, Li J, Nowak G, Allard MA, Jochmans I, Jacskon K, Beltrame MC, van Reeven M, Iesari S, Cucchetti A, Sharma H, Staiger RD, Raptis DA, Petrowsky H, de Oliveira M, Hernandez-Alejandro R, Pinna AD, Lerut J, Polak WG, de Santibanes E, de Santibanes M, Cameron AM, Pirenne J, Cherqui D, Adam RA, Ericzon BG, Nashan B, Olthoff K, Shaked A, Chapman WC, Boudjema K, Soubrane O, Paugam-Burtz C, Greig PD, Grant DR, Carvalheiro A, Muiesan P, Dutkowski P, Puhan M, Clavien PA. Defining Benchmarks in Liver Transplantation: A Multicenter Outcome Analysis Determining Best Achievable Results. Ann Surg. 2018 Mar;267(3):419-425. doi: 10.1097/SLA.0000000000002477. PMID 28885508
- [Background] Dindo D, Demartines N, Clavien PA. Classification of surgical complications: a new proposal with evaluation in a cohort of 6336 patients and results of a survey. Ann Surg. 2004 Aug;240(2):205-13. doi: 10.1097/01.sla.0000133083.54934.ae. PMID 15273542
- [Background] Slankamenac K, Graf R, Barkun J, Puhan MA, Clavien PA. The comprehensive complication index: a novel continuous scale to measure surgical morbidity. Ann Surg. 2013 Jul;258(1):1-7. doi: 10.1097/SLA.0b013e318296c732. PMID 23728278
- [Derived] Gero D, Raptis DA, Vleeschouwers W, van Veldhuisen SL, Martin AS, Xiao Y, Galvao M, Giorgi M, Benois M, Espinoza F, Hollyman M, Lloyd A, Hosa H, Schmidt H, Garcia-Galocha JL, van de Vrande S, Chiappetta S, Menzo EL, Aboud CM, Luthy SG, Orchard P, Rothe S, Prager G, Pournaras DJ, Cohen R, Rosenthal R, Weiner R, Himpens J, Torres A, Higa K, Welbourn R, Berry M, Boza C, Iannelli A, Vithiananthan S, Ramos A, Olbers T, Sepulveda M, Hazebroek EJ, Dillemans B, Staiger RD, Puhan MA, Peterli R, Bueter M. Defining Global Benchmarks in Bariatric Surgery: A Retrospective Multicenter Analysis of Minimally Invasive Roux-en-Y Gastric Bypass and Sleeve Gastrectomy. Ann Surg. 2019 Nov;270(5):859-867. doi: 10.1097/SLA.0000000000003512. PMID 31592894
- See also: Related Info — http://bbenchmarks.org